CLINICAL TRIAL: NCT07188103
Title: Efficacy and Safety of Ivonescimab Combined With Short-Course Hypofractionated Radiotherapy as Second-Line Therapy for Locally Advanced/Metastatic Esophageal Squamous Cell Carcinoma: A Prospective, Single-Center, Single-Arm Phase II Clinical Study
Brief Title: Ivonescimab Plus Short-Course Hypofractionated Radiotherapy as Second-Line Therapy for Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025KY-296
Record Dates: First submitted 2025-07-23; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal cancer; Hypofractionated Radiotherapy; Ivonescimab
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ivonescimab+Radiotherapy (Experimental): Short-course hypofractionated radiotherapy was administered to progressive lesions after first-line treatment, with a prescribed dose of 20 Gy in 5 fractions (95% PTV). The monoclonal antibody was initiated within 1 week after completing the radiotherapy regimen, at a dose of 20 mg/kg. Ivonescimab was administered every three weeks until disease progression, intolerable toxicity, or patient refusal.
  Interventions: Drug: Ivonescimab+Radiotherapy

INTERVENTIONS:
Drug: Ivonescimab+Radiotherapy — Short-course hypofractionated radiotherapy was administered to progressive lesions after first-line treatment, with a prescribed dose of 20 Gy in 5 fractions (95% PTV). The monoclonal antibody was initiated within 1 week after completing the radiotherapy regimen, at a dose of 20 mg/kg. Ivonescimab was administered every three weeks until disease progression, intolerable toxicity, or patient refusal.

SUMMARY:
In the era of immunotherapy, the standard second-line treatment regimen for locally advanced/metastatic esophageal squamous cell carcinoma (ESCC) remains controversial. This prospective, single-center, single-arm phase II clinical study aims to evaluate the efficacy and safety of Ivonescimab combined with short-course hypofractionated radiotherapy as a second-line therapy for patients with locally advanced/metastatic ESCC. The study plans to enroll 37 patients who have failed first-line treatment, without grouping, all of whom will receive Ivonescimab combined with short-course hypofractionated radiotherapy. The primary endpoints are progression-free survival (PFS) and safety, while the secondary endpoints include overall survival (OS), duration of response (DOR), and objective response rate (ORR). The study duration is 2 years.

ELIGIBILITY:
Inclusion Criteria:

* a. Patients with histologically confirmed esophageal squamous cell carcinoma (ESCC) , aged 18-80 years;
* b. Unresectable locally advanced, postoperative recurrent, or metastatic ESCC that has progressed on or is intolerant to first-line systemic therapy. For patients who received definitive concurrent chemoradiotherapy (CCRT) , disease progression during or within 6 months post-treatment is considered first-line treatment failure;
* c. At least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) . All positive regional lymph nodes are counted as a single lesion, while non-regional metastatic lymph nodes are counted per station;
* d. Adequate major organ function, defined as:

  1. Hematology:

     1. Hemoglobin (Hb) ≥ 90 g/L
     2. White blood cell (WBC) count ≥ 1.5 × 10⁹/L
     3. Platelet count ≥ 60 × 10⁹/L
  2. Serum biochemistry:

     1. Albumin ≥ 25 g/L
     2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal (ULN)
     3. Total bilirubin ≤ 1.5 × ULN
     4. Serum creatinine ≤ 1.5 × ULN or creatinine clearance (CrCl) ≥ 60 mL/min
  3. Echocardiography:

Left ventricular ejection fraction (LVEF) ≥ 50% (lower limit of normal)

* e. Eastern Cooperative Oncology Group (ECOG) performance status: 0-2;
* f. Expected survival ≥ 3 months;
* g. Voluntarily enrolled, with signed informed consent, and willing to comply with study protocols and follow-up.

Exclusion Criteria:

* a. Patients with severe organ dysfunction, uncontrolled acute infection, or significant comorbidities;
* b. Patients with vertebral metastases accompanied by spinal cord compression symptoms;
* c. Patients with esophagotracheal or esophagomediastinal fistulas;
* d. Patients with uncontrolled pleural, pericardial, or pelvic effusions requiring repeated drainage;
* e. Patients with esophageal primary/metastatic lesions invading the heart or great vessels, as assessed by the responsible physician, with a risk of life-threatening hemorrhage;
* f. Patients with esophageal primary/metastatic lesions invading the trachea or bronchi, as assessed by the responsible physician, with a risk of esophagotracheal fistula;
* g. Patients not suitable for short-course hypofractionated radiotherapy, as evaluated by the responsible physician;
* h. Pregnant or lactating women;
* i. Patients with mental disorders, or those with a history of psychotropic drug abuse and unable to quit;
* j. Patients who have participated in other drug clinical trials within the past 4 weeks;
* k. Patients or their families who refuse to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of enrollment until the date of first documented progression (radiologic or clinical), assessed every 8 weeks up to 36 months
  progression free survival
Advese Events | Assessed every 8 weeks up to 36 months from the date of enrollment
  Advese Events

SECONDARY OUTCOMES:
OS | From date of enrollment until the date of death from any cause, assessed up to 36 months
  overall survival
ORR | From enrollment to the time of the second radiological evaluation
  Objective Response Rate
DOR | the period from the first assessment of Complete Response (CR) or Partial Response (PR) to the first occurrence of Progressive Disease (PD) or death.
  Duration of Response
DCR | From enrollment to the time of second radiological evaluation
  Disease Control Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provincal Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided
undecided